CLINICAL TRIAL: NCT03982719
Title: Randomized Controlled Trial Comparing the Effectiveness of Two Post-fasciectomy Rehabilitation Protocols Differing in Intensity and Implementation of Modalities in Patients With Dupuytren's Disease
Brief Title: Comparing the Effectiveness of Two Post-fasciectomy Rehabilitation Protocols in Patients With Dupuytren's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Véronique Flamand (Other)
Collaborators: CHU de Quebec-Universite Laval (Other); Centre Interdisciplinaire de Recherche en Réadaptation et Intégration Sociale (Other)
Responsible Party: Sponsor-Investigator, Véronique Flamand, Assistant Professor and Researcher, Laval University
Organization: Laval University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dupuytren2019-4462
Record Dates: First submitted 2019-06-07; First posted 2019-06-11 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Dupuytren Contracture
Keywords: Dupuytren's disease; rehabilitation; fasciectomy; hand therapy
MeSH Terms: conditions — Dupuytren Contracture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief protocol (Experimental): 4 intervention sessions with the occupational therapist of 30 minutes duration.
  Interventions: Other: Brief protocol
- Intense Protocol (Active Comparator): 6 intervention sessions with the occupational therapist of 60 minutes duration.
  Interventions: Other: Intense protocol

INTERVENTIONS:
Other: Brief protocol — This protocol consists of 4 intervention sessions with an occupational therapist specialized in hand therapy that will occur at 0-3 days, 2 weeks, 4 weeks and 8 weeks post-fasciectomy. The occupational therapist will give recommendations about the management of swelling, wound care and functional recovery. An home exercises program will be given to the participant. The occupational therapist will make an extension splint that should be worn at night for the 3 months following surgery.
  Arms: Brief protocol
Other: Intense protocol — This protocol consists of 6 intervention sessions with an occupational therapist specialized in hand therapy that will occur at 0-3 days, 2 weeks, 3 weeks, 4 weeks, 6 weeks and 8 weeks after surgery. The occupational therapist will give recommendations about the management of swelling, wound care and functional recovery. An home exercises program will be given to the participant. The occupational therapist will make an extension splint that should be worn at night for the 3 months following surgery. Also, exercises will be performed by the patient under the supervision of the occupational therapist (supervised exercises) in each session except the first one at 0-3 days after surgery.
  Arms: Intense Protocol

SUMMARY:
Dupuytren's disease can cause physical impairments that lead to reduced functional performance in personal care, work-related and leisure activities. The prevalence of Dupuytren's disease increases with age. A meta-analysis completed in 2014 by Lanting and al. estimated the its prevalence in western countries at 12% among people aged 55 years and over and at 29% among individuals aged 75 and over. The fasciectomy is the most current surgical procedure to reduce the flexion contracture occurring in this disease. Studies confirm the relevance of post-operative rehabilitation after fasciectomy. This rehabilitation is usually conducted by hand therapists who are mostly occupational therapists. However, the required duration and frequency of interventions and exercises for the post-op rehabilitation are not clearly described in the literature. In fact, the guidelines that are currently available recommend a total duration between 16 and 75 hours, which is highly variable. Also, the need to include supervised exercises by the occupational therapist is not specified. The main goal of this study is to compare two post-fasciectomy rehabilitation protocols to determine the influence of protocols intensity on motor and functional outcomes in people with Dupuytren's disease. The hypothesis is that the protocol involving a higher intensity will lead to better motor and functional improvements. The secondary goal of this study is to explore the link between the total time that the person has done the recommended exercises (combination of supervised exercises and the home program) and motor/functional recovery. The hypothesis is that the relationship between the amount of time and the motor/functional improvements will not be linear, but will either be logarithmic toward a plateau of recovery.

A randomized controlled trial will be realized. 40 participants will be randomly assigned to one of the two rehabilitation protocols. Each participant will be evaluated at four times (initial evaluation, final evaluation and 2 follow-up evaluations). Data on motor and functional recovery will be collected.

DETAILED DESCRIPTION:
Dupuytren's disease can cause physical impairments that lead to reduced functional performance in personal care, work-related and leisure activities. The prevalence of Dupuytren's disease increases with age. A meta-analysis completed in 2014 by Lanting and al. estimated the its prevalence in western countries at 12% among people aged 55 years and over and at 29% among individuals aged 75 and over. The fasciectomy is the most current surgical procedure to reduce the flexion contracture occurring in this disease. Studies confirm the relevance of post-operative rehabilitation after fasciectomy. This rehabilitation is usually conducted by hand therapists who are mostly occupational therapists. However, the required duration and frequency of interventions and exercises for the post-op rehabilitation are not clearly described in the literature. In fact, the guidelines that are currently available recommend a total duration between 16 and 75 hours, which is highly variable. Also, the need to include supervised exercises by the occupational therapist is not specified. The main goal of this study is to compare two post-fasciectomy rehabilitation protocols to determine the influence of protocols intensity on motor and functional outcomes in people with Dupuytren's disease. The hypothesis is that the protocol involving a higher intensity will lead to better motor and functional improvements. The secondary goal of this study is to explore the link between the total time that the person has done the recommended exercises (combination of supervised exercises and the home program) and motor/functional recovery. The hypothesis is that the relationship between the amount of time and the motor/functional improvements will not be linear, but will either be logarithmic towards a plateau of recovery.

A randomized controlled trial will be realized. 40 participants will be randomly assigned to one of the two rehabilitation protocols. Each participant will be evaluated at four times (initial evaluation, final evaluation and 2 follow-up evaluations). The independent variable of this study is the intensity of the rehabilitation protocol (BRIEF or INTENSE). The primary dependent variable is the functional abilities to perform activities of daily living. The secondary dependent variables are the following : digits range of motion, pain, grip and pinch strengths, as well as tactile sensibility.

The BRIEF PROTOCOL consists of 4 intervention sessions with an occupational therapist specialized in hand therapy that will occur at 0-3 days, 2 weeks, 4 weeks and 8 weeks post-fasciectomy. The occupational therapist will give recommendations about the management of swelling, wound care and functional recovery. An home exercises program will be given to the participant. Finally, an extension splint that must be worn at night until the third month after surgery will be made at the first session. The INTENSE PROTOCOL consists of 6 intervention sessions with an occupational therapist specialized in hand therapy that will occur at 0-3 days, 2 weeks, 3 weeks, 4 weeks, 6 weeks and 8 weeks after surgery. The occupational therapist will give recommendations about the management of swelling, wound care and functional recovery. An home exercises program will be given to the participant. An extension splint that must be worn at night until the third month after surgery will be made at the first session. Also, exercises will be performed by the patient under the supervision of the occupational therapist (supervised exercises) in each session except the first one at 0-3 days after surgery.

Statistical analyses will take into account the moderate size of our sample (n=40) and the independence of the two groups. Descriptive statistics and Shapiro-Wilk test will be used to evaluate if variables follow the normal distribution. If the normal distribution is confirmed, repeated measure ANOVA will be used to compare the 2 groups. If not, Mann-Whitney test will be used (non-parametric test). Pearson correlation coefficient (parametric) or Spearman correlation coefficient (non-parametric) will be used to analyze the relationships between variables (secondary aim of the study).

ELIGIBILITY:
Inclusion Criteria:

* To present Dupuytren's contracture to one or two digits of the same hand and at an important stage of Dupuytren's Disease before the surgery (PIP contracture of 45 degrees or more)
* Having had a fasciectomy to treat Dupuytren's Disease with per-op PIP contracture of 30 degrees or less.

Exclusion Criteria:

* Recurrence of Dupuytren's Disease
* To have or have had a complex regional pain syndrome
* To present a health condition that could affect cognitive functions (dementia, neuro-cognitive disorders)
* To have a diagnosis of diabetes

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change from first evaluation on the Michigan Hand Questionnaire at 2, 3 and 6 months | 0-3 days, 2 months, 3 months and 6 months after surgery
  Patient-reported questionnaire that evaluates function and quality of life in patients with hand disorders. There are 37 items divided into 6 subscales (1)overall hand function, (2)activities of daily living, (3)pain, (4)work performance, (5)aesthetics and (6)patient's satisfaction with hand function). (Total score between 0-100, rating scale from 1 to 5)
Change from first evaluation on the Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) outcome measure at 2, 3 and 6 months | 0-3 days, 2 months, 3 months and 6 months after surgery
  Patient-reported questionnaire that evaluates 11 items on symptoms and functional impairments related to musculoskeletal disorders of the upper limb. (Total score between 0-100, rating scale from 1 to 5)
Change from first evaluation on the Sollerman Test at 2, 3 and 6 months | 2 months and 6 months after surgery
  A standardized hand function assessment based on seven of the eight most common hand grips that consists of 20 activities of daily living. (Total score between 0-80, rating scale 0 to 4).

SECONDARY OUTCOMES:
Range of motion assessed by Rolyan digital goniometer | 0-3 days, 2 months, 3 months and 6 months after surgery
  Range of motion of the affected digits assessed by Rolyan digital goniometer (data scope -30° to 120°, accuracy of 2°)
Pain measured using the Visual Analogue Scale | 0-3 days, 2 months, 3 months and 6 months after surgery
  Responders specify their level of pain by indicating a position along a continuous line between two end-points. One end (corresponding to score 0) represents the absence of pain, and the other end (corresponding to score 100) represents the worst pain that the person can imagine. (Thus the minimum score is 0, and the maximum score is 100. There are no sub-scales. 0 represents the absence of pain, and higher values represent more pain.)
Grip strength | 2 months, 3 months and 6 months after surgery
  JAMAR dynamometer (data scope 0-80 kg, accuracy of 2 kg)
Pinch strength | 2 months, 3 months and 6 months after surgery
  B&L pinch gauge (data scope 0-30 pounds, accuracy of 1 pound)
Tactile sensibility | 2 months, 3 months and 6 months after surgery
  Semmes-Weinstein monofilaments

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Flamand, PhD, Principal Investigator — Center for Interdisciplinary Research in Rehabilitation and Social Integration
Locations (1):
- CHU de Québec, Québec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ball C, Pratt AL, Nanchahal J. Optimal functional outcome measures for assessing treatment for Dupuytren's disease: a systematic review and recommendations for future practice. BMC Musculoskelet Disord. 2013 Apr 10;14:131. doi: 10.1186/1471-2474-14-131. PMID 23575442
- [Background] Bayat A, McGrouther DA. Management of Dupuytren's disease--clear advice for an elusive condition. Ann R Coll Surg Engl. 2006 Jan;88(1):3-8. doi: 10.1308/003588406X83104. PMID 16460628
- [Background] Bell-Krotoski JA, Fess EE, Figarola JH, Hiltz D. Threshold detection and Semmes-Weinstein monofilaments. J Hand Ther. 1995 Apr-Jun;8(2):155-62. doi: 10.1016/s0894-1130(12)80314-0. PMID 7550627
- [Background] Budd HR, Larson D, Chojnowski A, Shepstone L. The QuickDASH score: a patient-reported outcome measure for Dupuytren's surgery. J Hand Ther. 2011 Jan-Mar;24(1):15-20; quiz 21. doi: 10.1016/j.jht.2010.08.006. Epub 2010 Nov 24. PMID 21106346
- [Background] Desai SS, Hentz VR. The treatment of Dupuytren disease. J Hand Surg Am. 2011 May;36(5):936-42. doi: 10.1016/j.jhsa.2011.03.002. PMID 21527148
- [Background] Efanov JI, Shine JJ, Darwich R, Besner Morin C, Arsenault J, Harris PG, Danino AM, Izadpanah A. French translation and cross-cultural adaptation of the Michigan Hand Outcomes Questionnaire and the Brief Michigan Hand Outcomes Questionnaire. Hand Surg Rehabil. 2018 Apr;37(2):86-90. doi: 10.1016/j.hansur.2017.12.003. Epub 2018 Jan 17. PMID 29373241
- [Background] Huskisson EC. Measurement of pain. Lancet. 1974 Nov 9;2(7889):1127-31. doi: 10.1016/s0140-6736(74)90884-8. No abstract available. PMID 4139420
- [Background] Huisstede BMA, Hoogvliet P, Coert JH, Friden J; European HANDGUIDE Group. Dupuytren disease: European hand surgeons, hand therapists, and physical medicine and rehabilitation physicians agree on a multidisciplinary treatment guideline: results from the HANDGUIDE study. Plast Reconstr Surg. 2013 Dec;132(6):964e-976e. doi: 10.1097/01.prs.0000434410.40217.23. PMID 24281643
- [Background] Lanting R, Broekstra DC, Werker PMN, van den Heuvel ER. A systematic review and meta-analysis on the prevalence of Dupuytren disease in the general population of Western countries. Plast Reconstr Surg. 2014 Mar;133(3):593-603. doi: 10.1097/01.prs.0000438455.37604.0f. PMID 24263394
- [Background] Lewis E, Fors L, Tharion WJ. Interrater and intrarater reliability of finger goniometric measurements. Am J Occup Ther. 2010 Jul-Aug;64(4):555-61. doi: 10.5014/ajot.2010.09028. PMID 20825126
- [Background] Mathiowetz V, Weber K, Volland G, Kashman N. Reliability and validity of grip and pinch strength evaluations. J Hand Surg Am. 1984 Mar;9(2):222-6. doi: 10.1016/s0363-5023(84)80146-x. PMID 6715829
- [Background] Melchior H, Vatine JJ, Weiss PL. Is there a relationship between light touch-pressure sensation and functional hand ability? Disabil Rehabil. 2007 Apr 15;29(7):567-75. doi: 10.1080/09638280600902547. PMID 17453977
- [Background] Sollerman C, Ejeskar A. Sollerman hand function test. A standardised method and its use in tetraplegic patients. Scand J Plast Reconstr Surg Hand Surg. 1995 Jun;29(2):167-76. doi: 10.3109/02844319509034334. PMID 7569815
- [Background] Sweet S, Blackmore S. Surgical and therapy update on the management of Dupuytren's disease. J Hand Ther. 2014 Apr-Jun;27(2):77-83; quiz 84. doi: 10.1016/j.jht.2013.10.006. Epub 2013 Nov 5. PMID 24388681
- [Background] Wilburn J, McKenna SP, Perry-Hinsley D, Bayat A. The impact of Dupuytren disease on patient activity and quality of life. J Hand Surg Am. 2013 Jun;38(6):1209-14. doi: 10.1016/j.jhsa.2013.03.036. PMID 23707018